CLINICAL TRIAL: NCT03995446
Title: Low-level Laser Acupuncture Reduces Postoperative Pain and Morphine-related Side Effects in Patients With Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Low-level Laser Acupuncture Reduces Postoperative Pain and Morphine-related Side Effects in Patients With Total Knee Arthroplasty:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-02-007BCF
Record Dates: First submitted 2019-05-19; First posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Low-level Laser Acupuncture in Patients With Total Knee Arthroplasty
Keywords: Acupuncture points, low-level laser, postoperative pain, total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-level laser therapy (Experimental): 808nM wavelength, power density of 300mW
  Interventions: Device: low-level laser
- Sham laser acupuncture treatment (Sham Comparator): received the same manner except for joule.
  Interventions: Device: Sham laser

INTERVENTIONS:
Device: low-level laser — low level laser emission on specific acupuncture points
  Arms: low-level laser therapy
Device: Sham laser — Sham laser
  Arms: Sham laser acupuncture treatment

SUMMARY:
Total knee arthroplasty is a common and effective surgical procedure for patients with end-stage knee osteoarthritis, and wound pain is still a problem for many of the patients.

DETAILED DESCRIPTION:
Therefore, the purpose of this study was to apply low level laser therapy Measured variables included postoperative pain intensity, patient-controlled analgesia requirements, side effects caused by morphine, knee stiffness and wound pain in the daily activities of patients undergoing total knee arthroplasty. Data were collected between April 2018 and January 2019. Eighty-two knee osteoarthritis patients receiving total knee arthroplasty were recruited from one hospital and randomly, equally assigned to the laser acupuncture or control group. The LA group received the low-level laser therapy with 3 joules at each acupuncture point at Hour 2, Hour 6, Hour 10, Hour 24, Hour 48, and Hour 72 after surgery; whereas the control group received the same manner except for joule.

ELIGIBILITY:
Inclusion Criteria:

* age 60 years or older
* American Sociological Association (ASA) class I-III
* spinal anesthesia, consent to patient-controlled analgesia (PCA) and peripheral nerve block (PNB)
* return to the ward directly from the anesthesia recovery room.

Exclusion Criteria:

* cutaneous lesions at the application sites
* use of taking immunosuppressive agents
* received intra-articular steroid treatment
* opiate dependence
* sensitive to light
* epilepsy
* clinically significant cardiovascular diseases
* cancer
* systemic lupus erythematosus.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-04-21 (Actual)

PRIMARY OUTCOMES:
The Numerical Rating Scale (NRS) | the first 72 hours after the surgery
  NRS was assessed pain intensity, ranging from 0 (no pain) to 10 (worst pain imaginable).higher scores, higher pain.
Brief Pain Inventory (BPI) | the first 72 hours after the surgery
  The patients answered or pointed their pain on 0-to-10 scales (0=no pain, 10=extreme pain) at the time of responding to the BPI(current pain), and also at the items of "the most severe pain", "the least pain", and "the average pain" in the last 24 hours. Using the BPI, patients were also asked to rate pain-related interference in daily activities, including general activity, mood, walking ability, normal work, relations with other people, sleeping, and enjoyment of life. The anchor points, in each items of interference scale, were 11-point NRSs (0=no interference, 10=interferes completely).

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veteran General Hospital : Taipei City, Taiwan 11217, R.O.C., Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang CH, Yeh ML, Chen FP, Wu D. Low-level laser acupuncture reduces postoperative pain and morphine consumption in older patients with total knee arthroplasty: A randomized placebo-controlled trial. J Integr Med. 2022 Jul;20(4):321-328. doi: 10.1016/j.joim.2022.04.002. Epub 2022 Apr 9. PMID 35459599